CLINICAL TRIAL: NCT07037628
Title: Investigating the Impact of Spinal Cord Electrical Stimulation Combined With Individualized Physical Therapy on Lower Extremity Function in Patients With Spinal Cord Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Lian-Cing Yan, MSPT (Other)
Responsible Party: Sponsor-Investigator, Lian-Cing Yan, MSPT, Physical therapist, Hualien Tzu Chi General Hospital
Organization: Hualien Tzu Chi General Hospital (Other)
Other Study IDs: IRB114-106-B
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injury; Spinal Cord Injury Thoracic; Spinal Cord Injury/Damage; Spinal Cord Injury T1-L2; Spinal Cord Stimulation (SCS); Spinal Cord Stimulation; Epidural Electrical Stimulation
Keywords: ASIA B; ASIA C; ASIA D; ASIA A
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Spinal cord stimulation (SCS) combined with one-on-one physical therapy
- Control group: One-on-one physical therapy only

SUMMARY:
This study aims to understand the differences in the effects of two rehabilitation approaches on lower limb function recovery in patients with spinal cord injuries:

1. Spinal cord stimulation (SCS) combined with one-on-one physical therapy
2. One-on-one physical therapy alone

DETAILED DESCRIPTION:
This study adopts a prospective controlled design to observe and explore the effect of SCS combined with one-on-one physical therapy on the recovery of lower limb function in patients with spinal cord injury. The aims is to collect clinical practice data and provide reference for future related treatment strategies and care, hoping to increase the treatment options for rehabilitation of patients with spinal cord injury and improve their functional performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 70 years.
* Diagnosed with spinal cord injury, classified as ASIA Grade A-D.
* Neurological level of injury between T1 and L2.
* Spinal cord injury has stabilized (for at least 3 months).
* Currently receiving standard treatment at Hualien Tzu Chi Hospital and referred by a neurosurgeon or orthopedic surgeon to receive spinal cord stimulation (SCS) and/or individualized physical therapy.
* Capable of participating in one-on-one physical therapy sessions 3 to 5 times per week, and assessed by the medical team as able to complete at least a 3 weeks course of treatment.
* Fully conscious, able to understand the study information, and willing to sign the consent form and participate in the full assessment process.

Exclusion Criteria:

* Individuals with severe brain injury, neurodegenerative diseases, or other major neurological disorders.
* Those with severe fractures, joint contractures, or conditions preventing participation in lower limb training.
* Individuals with a cardiac pacemaker or who are pregnant.
* Those unable to comply with the treatment or assessment procedures.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Currently receiving standard treatment at Hualien Tzu Chi Hospital and referred by a neurosurgeon or orthopedic surgeon for spinal cord stimulation (SCS) and/or individualized physical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Impairment Scale | Experimental group:To measure assessing change between pre-implant and one month after implant. Control group:To measure assessing change between Day 1 and one month after physical therapy.
  -AIS A (Complete): S4-S5 have no sensory and motor function.
  -AIS B (Sensory Incomplete): S4-S5 have sensory function (light touch or pinprick sensation or deep anal pressure sensation), but no motor function.
  And the motor function score of more than three levels below the injury plane is 0.
  -AIS C (Motor Incomplete): S4-S5 have motor function (voluntary anal sphincter contraction), or the sacral ganglion has sensory function and more than half of the key muscle groups below the injury plane have a strength of less than 3 points.
  -AIS D (Motor Incomplete): The muscle strength of at least half of the key muscle groups below the injury plane is greater than or equal to 3 points.
  -AIS E (Normal): Both sensory and motor functions are tested normal.
Modified Ashworth Scale (MAS) | Experimental group:To measure assessing change between pre-implant and one month after implant. Control group:To measure assessing change between Day 1 and one month after physical therapy.
  Grade judgment:
  * 0 points: No increase in muscle tension.
  * 1 point: Slight increase in muscle tension at the end of the joint range of motion, manifested as a sudden jam and immediate relaxation.
  * 1+ points: Slight increase in muscle tension in less than half of the joint range of motion, followed by minimal resistance in the remaining range of motion.
  * 2 points: Significant increase in muscle tension in most of the joint range of motion, but the joint can still be moved easily.
  * 3 points: Significant increase in muscle tension, passive movement becomes difficult.
  * 4 points: The joint becomes stiff in flexion or extension and cannot be moved passively.
Handheld Dynamometer | Experimental group:To measure assessing change between pre-implant and one month after implant. Control group:To measure assessing change between Day 1 and one month after physical therapy.
  Force application method: The assessor instructs the patient to resist with all his strength, and the assessor gradually applies force until the patient is unable to resist and collapses, and the maximum force value is recorded.
  Data recording: 3 measurements are performed and the average value is taken. The unit of force is pounds (lbs).
Spinal Cord Independence Measure (SCIM III) | Experimental group:To measure assessing change between pre-implant and one month after implant. Control group:To measure assessing change between Day 1 and one month after physical therapy.
  Grade determination (scoring): Total score 0-100 points.
  - Scoring principle: The higher the score, the better the patient's independence. The scoring criteria for each item are different.
  The core concept is to give points based on the degree of assistance required by the patient when actually performing the task.
  * High score: Completely independent, or only requires a small amount of assistive devices.
  * Medium score: Partial assistance is required (for example: verbal prompts, others preparing items, a small amount of physical assistance).
  * Low score: A lot of assistance is required or completely dependent on others.
World Health Organization Quality-of-Life Scale | Experimental group:To measure assessing change between pre-implant and one month after implant. Control group:To measure assessing change between Day 1 and one month after physical therapy.
  Grade determination (0-20): A hierarchical scale from 0 to 20, with higher numbers representing better walking function and lower dependence.
  * Grade 0: The patient cannot stand or walk.
  * Grade 1-5: Requires physical assistance from 2 therapists and may use different types of braces. The higher the grade, the fewer braces are needed.
  * Grade 6-8: Requires physical assistance from 1 therapist and may use different types of braces or walkers.
  * Grade 9-12: No assistance from others, but requires a walker and may use different types of braces.
  * Grade 13-16: No assistance from others, but requires the use of two crutches and may use different types of braces.
  * Grade 17-19: No assistance from others, but requires the use of a single crutch or cane and may use a brace.
  * Grade 20: Walk 10 meters on flat ground without any physical assistance, braces or assistive devices.
Walking Index for Spinal Cord Injury (WISCI II) | Experimental group:To measure assessing change between pre-implant and one month after implant. Control group:To measure assessing change between Day 1 and one month after physical therapy.
  Grade determination (0-20): A hierarchical scale from 0 to 20, with higher numbers representing better walking function and lower dependence.
  * Grade 0: The patient cannot stand or walk.
  * Grade 1-5: Requires physical assistance from 2 therapists and may use different types of braces. The higher the grade, the fewer braces are needed.
  * Grade 6-8: Requires physical assistance from 1 therapist and may use different types of braces or walkers.
  * Grade 9-12: No assistance from others, but requires a walker and may use different types of braces.
  * Grade 13-16: No assistance from others, but requires the use of two crutches and may use different types of braces.
  * Grade 17-19: No assistance from others, but requires the use of a single crutch or cane and may use a brace.
  * Grade 20: Walk 10 meters on flat ground without any physical assistance, braces or assistive devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Buddhist Tzu Chi Medical Foundation Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No